CLINICAL TRIAL: NCT01583933
Title: PHASE 3 STUDY OF THE EFFECTIVITY OF TWO RETAINERS IN THE DENTAL AND OCCLUSAL STABILITY
Brief Title: Essix Retainer vs Hawley Retainer
Acronym: retainer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CES University (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Angela Maria Segura Cardona, Research, CES University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFHA-02
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Dental and Occlusal Stability
Keywords: Dental stability; Occlusal stability; Retainers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Essix retainer (Experimental)
  Interventions: Device: Essix retainer
- Hawley retainer (Active Comparator): Hawley retainer is a device composed of an acrylic base with built-in hooks and a labial arch wire 0.022 "x0.036" and attached to the teeth. Its metal component consists of two adams hooks positioned from the first permanent molar right to left, a labial bow that progresses from lingual superface to distal of canine to integrate with the acrylic base.
  Interventions: Device: Hawley retainer

INTERVENTIONS:
Device: Essix retainer — The essix retainer is made in a thermoforming copolyester 0.75mm (0.30 ", it processed gives a thickness of 0.015" approximately. Retainer will be used molar to molar. subjects in this arm will have this retainer for 24 hours a day for 6 months, they won´t have this device for food intake.
  Arms: Essix retainer
Device: Hawley retainer — subjects in this arm will have the retainer for 24 hours a day for 6 months. During food intake they won´t have this device.
  Arms: Hawley retainer

SUMMARY:
There are several factors involved in the decision and the retention plan, such as occlusion, patient age, etiology of malocclusion, the speed of the correction, the length of the cusps and health of the tissues involved, relationships inclined planes, size of the arches, harmony of the arches, muscle pressure, interdental proximal contact, cell metabolism and atmospheric pressure. Given these concepts, we need to find grounds to enable decision making with respect to the retainer that offers the best features of containment and stability.

DETAILED DESCRIPTION:
This study aims to assess the stability of tooth position and occlusal retention during treatment with two types of retainers, Essix type retainer and the retainer plate type Hawley in individuals who have completed their growth ending orthodontic treatment at the Faculty of Dentistry University of Antioquia and CES University Medellín

ELIGIBILITY:
Inclusion Criteria:

* Patients who have stabilized their growth between 16 and 40 who have completed orthodontic treatment and initiate retention treatment
* Who have agreed to participate in the study if elected and to sign informed consent
* Residing in the metropolitan area of Medellin and have the opportunity to attend recall appointments

Exclusion Criteria:

* Periodontal status deteriorated
* missing teeth
* Cleft lip and palate
* History of orthognathic surgery
* History of dental or skeletal open bite
* Presence of some habit oral tongue thrusting, mouth breathing, thumb sucking even after termination of orthodontic treatment

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Dental stability | Up to 6 months
  Dental stability will be assessed like this, models: rotation of central and lateral incisor, canine, first and second premolar, first molar on each side and each arch; and cephalometric analysis: SN-upper central incisive, FK-upper central incisive, palate plane-upper central incisive, interincisal angle, mandibular plane-lower central incisive; vertical distances: palate plane-upper central incisive, palate plane-first upper molar, mandibular plane-lower central incisive, mandibular plane-first lower molar; horizontal distances: A-Pogonion upper and lower central incisive.

SECONDARY OUTCOMES:
Occlusal stability | Up to 6 months
  Occlusal stability will be measured at the beginning and end of study through clinic exam and study models.
  Clinic exam: canine relations right and left, molar relations left and right, overjet, overbite, presence of anterior open bite, presence of posterior open bite.
  Models: upper and lower arch, upper and lower intercanine distance, upper and lower distance interpremolar, upper and lower intermolar distance.

CONTACTS AND LOCATIONS:
Locations (1):
- CES University, Medellín, Antioquia, Colombia